CLINICAL TRIAL: NCT01441583
Title: Ingenio Device Algorithm Study
Acronym: IVORY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-CL-07202011-B-H
Record Dates: First submitted 2011-09-26; First posted 2011-09-27 (Estimated); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Sinus Node Disease; AV Block; Heart Failure
Keywords: pacemaker, CRT-P, auto threshold
MeSH Terms: conditions — Sick Sinus Syndrome; Atrioventricular Block; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pacemaker - RYTHMIQ Off at Pre-discharge, On at 1-Month (Active Comparator): For the RYTHMIQ endpoint only, subjects implanted with a pacemaker will be randomized. Those randomized to RYTHMIQ Off at Pre-Discharge will have RYTHMIQ programmed Off until their 1-month follow up, when they will be crossed over to RYTHMIQ On until their 3-month follow up.
  Interventions: Device: RAAT; Device: RYTHMIQ
- Pacemaker - RYTHMIQ On at Pre-Discharge, Off at 1-Month (Active Comparator): For the RYTHMIQ endpoint only, subjects implanted with a pacemaker will be randomized. Those randomized to RYTHMIQ On at Pre-Discharge will have RYTHMIQ programmed On until their 1-month follow up, when they will be crossed over to RYTHMIQ Off until their 3-month follow up.
  Interventions: Device: RAAT; Device: RYTHMIQ
- CRT-P (Experimental): CRT-P devices were not involved in RYTHMIQ endpoint evaluation, only RAAT.
  Interventions: Device: RAAT

INTERVENTIONS:
Device: RAAT — For Pacemaker and CRT-P: Right Atrial Automatic Threshold (RAAT)
Device: RYTHMIQ — For pacemakers only: RYTHMIQ RYTHMIQ randomized to on at pre-discharge or at 1-month, depending on assignment
  Arms: Pacemaker - RYTHMIQ Off at Pre-discharge, On at 1-Month; Pacemaker - RYTHMIQ On at Pre-Discharge, Off at 1-Month

SUMMARY:
The purpose of the IVORY Study is to gather data to support global submissions/approvals for some models of the Ingenio device family.

DETAILED DESCRIPTION:
IVORY is a prospective, multi-center, randomized within-patient, single-blinded study to gather data to support Right Atrial Auto Threshold and RYTHMIQ

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are willing and capable of providing informed consent to undergo a device implant and to participate in all testing associated with this clinical study;
* Subjects whose age is 18 or above, or of legal age to give informed consent specific to national law;
* Subjects indicated for a dual chamber pacemaker or a CRT-P device according to class I or class II indications of the standard ESC or ACC / AHA implant guidelines;
* Subjects who are planned to be implanted with all leads intended for a specific device type (dual chamber pacemaker: atrial and right ventricular lead, CRT-P: atrial, right and left ventricular lead) or are already implanted with such leads;
* Subjects who receive or are implanted with a bipolar atrial lead.

Exclusion Criteria:

* Women of childbearing potential who are or might be pregnant at the time of the study (method of assessment upon physician's discretion);
* Enrolled in any other concurrent study, with the exception of local mandatory governmental registries and observational studies/registries that are not in conflict or affect
* Schedule of procedures for IVORY (i.e. should not cause additional or missed visits);
* Programming of devices for IVORY per CIP;
* IVORY outcome (i.e. involve medications that could affect the heart rate of the subject);
* Conduct of IVORY per GCP / ISO 14 155:2011 / local regulations.
* Subjects who live at such a distance from the clinic that travels for FU visits at a study center would be unusually difficult or burdensome for the subject;
* Inability or refusal to comply with the FU schedule;
* A life expectancy of less than 12 months, per physician discretion;
* Subjects who are planned to be programmed to a pacing mode other than DDD / DDDR during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-10; Primary Completion 2012-06 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy S Gardner, MD, Principal Investigator — Golden Jubilee National Hospital; Jens Goetzke, Dipl.-Ing. (FH), Study Director — Boston Scientific Corporation
Locations (21):
- Austria (2):
  - Wilhelminenspital, Vienna
  - Landesklinikum Wiener Neustadt, Wiener Neustadt
- Clinique Universitaires Saint Luc, Brussels, Belgium
- Denmark (2):
  - Rigshospitalet Copenhagen, Copenhagen
  - Gentofte University Hospital, Hellerup
- France (2):
  - NCN Nouvelles Cliniques Nantaises, Nantes
  - Clinique Saint-Hilaire Rouen, Rouen
- Germany (2):
  - Krankenhaus Neu Bethlehem, Göttingen
  - Heinrich Braun Krankenhaus, Zwickau
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Italy (2):
  - Azienda Ospedaliera Mater Domini Policlinico Universitario, Catanzaro, CZ
  - Policlinico Casilino, Roma, RM
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- Netherlands (2):
  - Amphia Ziekenhuis, Breda
  - Rijnland Ziekenhuis, Leiderdorp
- Spain (2):
  - Hospital Clinico Y Provincial, Barcelona
  - Clinica Universitaria de Navarra, Pamplona
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska Hospital, Stockholm
- United Kingdom (2):
  - Golden Jubilee National Hospital, Clydebank
  - Northern General Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the general patient population indicated for a dual chamber pacemaker or cardiac resynchronization therapy pacemaker implantation at 15 study centers. First enrollment date was in October 2011 and the last subject was enrolled in March 2012.
Pre-assignment Details: Of 139 subjects, 132 were implanted with a study device. Of those subjects who were not implanted with a study device 4 signed informed consent, met eligibility criteria and had anesthesia administered in preparation for the surgical procedure but did not receive a study device (classified as 'Attempt') and 3 signed the informed consent, met eligibility criteria but did not undergo an implant (classified as an 'Intent').
Groups:
- RYTHMIQ Off at Pre-discharge, On at 1-Month: Pacemaker - RYTHMIQ Off at Pre-discharge, On at 1-Month
- RYTHMIQ On at Pre-Discharge, Off at 1-Month: Pacemaker -RYTHMIQ On at Pre-Discharge, Off at 1-Month
- CRT-P: All CRT-P implanted subjects
Period: Overall Study
Arm/Group | RYTHMIQ Off at Pre-discharge, On at 1-Month | RYTHMIQ On at Pre-Discharge, Off at 1-Month | CRT-P
Started | 50 | 50 | 36
Completed | 48 | 49 | 27
Not Completed | 2 | 1 | 9
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Death | 1 | 0 | 4
Not completed — Underwent anaesthesia, but not finally implanted | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Baseline Analysis Population includes all implanted subjects (n=132) as well as 4 attempted CRT-P subjects that could not be successfully implanted but underwent anesthesia. Total baseline population is therefore n=136.
Groups:
- Pacemaker: Subjects receiving a pacemaker study device (implanted or attempted)
- CRT-P: Subjects receiving a CRT-P study device (implanted or attempted)
- Total: Total of all reporting groups
Arm/Group | Pacemaker | CRT-P | Total
Number analyzed (Participants) | 100 | 36 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.3 (10.9) | 72.7 (9.5) | 73.2 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 28 | 88
  Male | 40 | 8 | 48
Pacemaker Indication [Count of Participants; unit: Participants] — Not applicable for CRT-P device category Population: Pacemaker indications are not applicable for CRT-P device category, hence it was not analyzed.
  Participants
    AV Block: number analyzed (Participants) | 100 | 0 | 100
    AV Block | 56 | 0 | 56
    Sinus Node Dysfunction: number analyzed (Participants) | 100 | 0 | 100
    Sinus Node Dysfunction | 37 | 0 | 37
    Other Block (i.e. Chronic Bifascicular Block): number analyzed (Participants) | 100 | 0 | 100
    Other Block (i.e. Chronic Bifascicular Block) | 5 | 0 | 5
    Hypersensitive Carotid Sinus Syndrome: number analyzed (Participants) | 100 | 0 | 100
    Hypersensitive Carotid Sinus Syndrome | 1 | 0 | 1
    Brady-Tachy Syndrome: number analyzed (Participants) | 100 | 0 | 100
    Brady-Tachy Syndrome | 1 | 0 | 1
CRT-P Indication [Count of Participants; unit: Participants] — Class I indication (ind.) for CRT-P device, defined by Left Ventricular Ejection Fraction (EF) = ≤ 35%, sinus rhythm, NYHA Class III, or ambulatory NYHA Class IV, QRS width (QRS) of ≥ 120 ms and optimal heart failure drug therapy (OPT). Recommended ind.
  Class IIa, defined by EF ≤ 35%, NYHA Class III, or ambulatory NYHA Class IV, OPT, frequent dependence on ventricular pacing. Ind. should be considered.
  Class IIb, defined by EF ≤ 35%, NYHA Class I or II, OPT, device implant with anticipated frequent ventricular pacing. Ind. can be considered.
  Not applicable for pacemaker device category. Population: CRT-P indications are not applicable for pacemaker device category, hence it was not analyzed.
  Participants
    Class I - EF ≤ 35%, sinus rhythm, NYHA Class III, or ambulatory NYHA Class IV, QRS ≥ 120 ms, OPT: number analyzed (Participants) | 0 | 36 | 36
    Class I - EF ≤ 35%, sinus rhythm, NYHA Class III, or ambulatory NYHA Class IV, QRS ≥ 120 ms, OPT | 0 | 19 | 19
    Class IIa - EF ≤ 35%, NYHA Class III, or ambul. NYHA Class IV, OPT, freq. dependence on vent. pacing: number analyzed (Participants) | 0 | 36 | 36
    Class IIa - EF ≤ 35%, NYHA Class III, or ambul. NYHA Class IV, OPT, freq. dependence on vent. pacing | 0 | 4 | 4
    Class IIb - EF ≤ 35%, NYHA Class I or II, OPT, device implant with anticipated frequent vent. pacing: number analyzed (Participants) | 0 | 36 | 36
    Class IIb - EF ≤ 35%, NYHA Class I or II, OPT, device implant with anticipated frequent vent. pacing | 0 | 5 | 5
    Replacement CRT-P device: number analyzed (Participants) | 0 | 36 | 36
    Replacement CRT-P device | 0 | 6 | 6
    Other: number analyzed (Participants) | 0 | 36 | 36
    Other | 0 | 2 | 2
NYHA Class [Count of Participants; unit: Participants] — New York Heart Association (NYHA) Classification places subjects into one of four categories based on their physical activity limitations with Class I = no limitations, Class II = Mild limitations, Class III = Moderate limitations and Class IV = Severe limitations.
  Participants
    I | 24 | 1 | 25
    II | 10 | 8 | 18
    III | 2 | 21 | 23
    IV | 0 | 3 | 3
    Not reported | 64 | 3 | 67
LVEF [Mean (Standard Deviation); unit: percent] — Population: Measure not reported for all subjects.
  percent
    number analyzed (Participants) | 43 | 33 | 76
    (all) | 55.7 (10.5) | 29.2 (8.4) | 44.1 (16.3)
QRS Duration [Mean (Standard Deviation); unit: ms] — Population: Measure not reported for all subjects.
  ms
    number analyzed (Participants) | 82 | 32 | 114
    (all) | 109 (33) | 158 (24) | 123 (38)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Measure not reported for all subjects.
  kg/m^2
    number analyzed (Participants) | 87 | 33 | 120
    (all) | 26.3 (4.1) | 27.2 (4.0) | 26.6 (4.1)
Body Surface Area [Mean (Standard Deviation); unit: m^2] — Population: Measure not reported for all subjects.
  m^2
    number analyzed (Participants) | 87 | 33 | 120
    (all) | 1.9 (0.3) | 1.9 (0.2) | 1.9 (0.2)
Concomitant Medications [Count of Participants; unit: Participants] — Subjects may contribute to more than one category.
  Participants
    ACE Inhibitor | 27 | 18 | 45
    Angiotensin Receptor Blocker | 26 | 16 | 42
    Diuretics | 26 | 27 | 53
    Sodium Channel Blockers - Class I | 3 | 0 | 3
    Beta Blockers - Class II | 26 | 26 | 52
    Potassium Channel Blockers - Class III | 4 | 3 | 7
    Calcium Channel Blockers - Class IV | 26 | 4 | 30
    Other Cardiovascular Medications | 60 | 29 | 89
Etiology [Count of Participants; unit: Participants]
  No Disease (age related) | 80 | 4 | 84
  Ischemic Cardiomyopathy | 10 | 17 | 27
  Idiopathic Cardiomyopathy | 3 | 12 | 15
  Valvular Cardiomyopathy | 4 | 3 | 7
  Congenital Heart Disease | 2 | 0 | 2
  Hypertrophic Cardiomyopathy | 1 | 0 | 1
Atrial Arrhythmias [Count of Participants; unit: Participants] — Subjects may contribute to more than one category
  Participants
    Paroxysmal Atrial Fibrillation | 18 | 8 | 26
    Atrial Tachycardia/Flutter | 7 | 3 | 10
    Persistent Atrial Fibrillation | 1 | 0 | 1
    Other Supraventricular Tachycardia | 3 | 0 | 3
    None | 72 | 26 | 98
Brady Arrhythmias: [Count of Participants; unit: Participants] — Subjects may contribute to more than one category
  Participants
    Sinus Node Dysfunction | 32 | 1 | 33
    3rd Degree AV Block - Intermittent | 21 | 3 | 24
    2nd Degree AV Block - Intermittent | 17 | 2 | 19
    3rd Degree AV Block - Permanent | 15 | 4 | 19
    1st Degree AV Block | 12 | 6 | 18
    Bradycardia | 14 | 2 | 16
    2nd Degree AV Block - Permanent | 10 | 0 | 10
    Sinus Arrest | 7 | 0 | 7
    Chronotropic Incompetence | 5 | 0 | 5
    None | 6 | 20 | 26
Cardiac Disease & Arrhythmia HistorY [Count of Participants; unit: Participants] — Subjects may contribute to more than one category
  Participants
    Hypertension | 64 | 12 | 76
    Diabetes | 23 | 11 | 34
    Heart Failure | 6 | 23 | 29
    Chronic Pulmonary Disease | 10 | 4 | 14
    Renal Disease | 5 | 6 | 11
    Other | 26 | 8 | 34
    None | 25 | 4 | 29

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Commanded Right Atrial Automatic Threshold (RAAT)
Description: Accuracy was evaluated by the proportion of tests resulting in an RAAT commanded threshold with |Manual unipolar threshold - commanded threshold| ≤ 0.5V. Subjects were allowed to contribute multiple paired datasets for this endpoint analysis, one set each from the 1-month and 3-month visits. Paired datasets from the 1-month and 3-month visits were pooled for purposes of endpoint analysis. A paired dataset consisted of the manual unipolar threshold and the commanded threshold obtained at a visit.
Time Frame: 3 months post implant
Population: Arms/Groups are only applicable for the outcome measure 'Secondary Outcome: RYTHMIQ - Median Relative Reduction of RV Pacing Percent (RVPP) for RYTHMIQ Programmed to ON vs. RYTHMIQ Programmed to OFF'.
  This outcome measure was analyzed only for the combined population. Analysis performed on subjects with paired datasets, each consisting of a commanded RAAT threshold and manual unipolar threshold collected at the 1- and 3-month visits.
Measure: Number (95% Confidence Interval); unit: percentage of accurate RAAT tests
Units Other Than Participants: Paired threshold tests
Groups:
- RAAT Commanded Threshold: Subjects with paired RAAT commanded threshold and manual unipolar threshold available
Arm/Group | RAAT Commanded Threshold
Number analyzed (Participants) | 132
Number analyzed (Paired threshold tests) | 190
percentage of accurate RAAT tests | 100 [96.8 to 100]

2. Primary Outcome: System-related Complication-free Rate
Description: Arms/Groups are only applicable for the outcome measure 'Secondary Outcome: RYTHMIQ - Median Relative Reduction of RV Pacing Percent (RVPP) for RYTHMIQ Programmed to ON vs. RYTHMIQ Programmed to OFF'.
  This outcome measure was analyzed only for the combined population and both pacemakers and CRT-P devices were pooled for the analysis. The analysis assesses the system-related complication (SRC) -free rate (excluding LV related events for CRT-P subjects) for subjects implanted or attempted to be implanted with a study device through the first 90 days following the implant procedure.
Time Frame: 90 days post-implant
Measure: Number (95% Confidence Interval); unit: percentage of subjects free from SRC
Groups:
- Implanted or Attempted: All subjects, who were implanted with a study device or attempted to be implanted with a study device.
Arm/Group | Implanted or Attempted
Number analyzed (Participants) | 136
percentage of subjects free from SRC | 87.5 [81.8 to 100]

3. Secondary Outcome: Accuracy of Ambulatory RAAT
Description: Arms/Groups are only applicable for the outcome measure 'Secondary Outcome: RYTHMIQ - Median Relative Reduction of RV Pacing Percent (RVPP) for RYTHMIQ Programmed to ON vs. RYTHMIQ Programmed to OFF'.
  This outcome measure was analyzed only for the combined population (pacemaker and CRT-P). Accuracy was evaluated by the proportion of tests resulting in an RAAT ambulatory threshold with |ambulatory threshold - commanded threshold| ≤ 1.0V. Subjects were allowed to contribute multiple paired datasets for this endpoint analysis, one set each from the 1-month and 3-month visits. Paired datasets from the 1-month and 3-month visits were pooled for purposes of endpoint analysis. A paired dataset consisted consisted of the ambulatory threshold obtained within 7 days prior to the visit and the commanded threshold obtained at the visit.
Time Frame: 3 months post-implant
Measure: Number (95% Confidence Interval); unit: Paired threshold tests
Units Other Than Participants: Paired threshold tests
Groups:
- Implanted: All subjects, who were implanted with a study device
Arm/Group | Implanted
Number analyzed (Participants) | 132
Number analyzed (Paired threshold tests) | 187
Paired threshold tests | 186 [182 to 187]

4. Secondary Outcome: Appropriate RAAT Test Outcome
Description: Arms/Groups are only applicable for the outcome measure 'Secondary Outcome: RYTHMIQ - Median Relative Reduction of RV Pacing Percent (RVPP) for RYTHMIQ Programmed to ON vs. RYTHMIQ Programmed to OFF'.
  This outcome measure was analyzed only for the combined population (pacemaker and CRT-P). Accuracy was evaluated by the proportion of tests with an appropriate commanded RAAT test outcome. An appropriate RAAT outcome consists of either a device-determined threshold or a code indicating that a threshold could not be determined and representing a condition that is beyond the control of the RAAT feature and could occur as well in manual threshold test, such as atrial fibrillation.
Time Frame: 3 months post-implant
Measure: Number (95% Confidence Interval); unit: percentage of approprite RAAT tests
Units Other Than Participants: threshold tests
Arm/Group | Implanted
Number analyzed (Participants) | 132
Number analyzed (threshold tests) | 242
percentage of approprite RAAT tests | 84.7 [80.4 to 100]

5. Secondary Outcome: RYTHMIQ - Median Relative Reduction of RV Pacing Percent (RVPP) for RYTHMIQ On at Pre-Discharge, Off at 1-Month vs. RYTHMIQ Off at Pre-discharge, On at 1-Month
Description: Chronic success is assessed by a median relative reduction of RV pacing percent (RVPP) for RYTHMIQ On at Pre-Discharge, Off at 1-Month vs. RYTHMIQ On at Pre-Discharge, Off at 1-Month. All patients received both RYTHMIQ programmed to ON and programmed to OFF in two consecutive periods, where the patient's programming allocation was randomized for the first period. Then a crossover to the alternate setting occurred for the second period once the end of the first period was reached.
Time Frame: 3 months post implant
Population: Pacemaker subjects with RYTHMIQ information available for both randomization periods.
Measure: Median (Full Range); unit: Percentage of RV pacing
Groups:
- Pacemaker Subjects Without Permanent 3° AV Block: Subjects receiving a pacemaker study device (implanted or attempted) except those with permanent 3° AV Block
Arm/Group | Pacemaker Subjects Without Permanent 3° AV Block
Number analyzed (Participants) | 84
Percentage of RV pacing
  RYTHMIQ On | 4 [0 to 100]
  RYTHMIQ Off | 98 [1 to 100]

6. Secondary Outcome: Percentage of RAAT Threshold Tests With Sufficient RAAT Pace Output Margin
Description: This outcome measure was analyzed only for the combined population (Pacemaker and CRT-P). The sufficient pacing output voltage that is able to capture the right atrium was evaluated by the proportion of Right Atrial Automatic Threshold (RAAT) tests with [RAAToutput ≥ (max(BP,UP) + δ )] where BP refers to the manual bipolar threshold, UP refers to the manual unipolar threshold, and δ refers to the safety margin of 0.5V. Subjects were allowed to contribute multiple paired datasets for this endpoint analysis, one set each from the 1-month and 3-month visits. Paired datasets from the 1-month and 3-month visits were pooled for purposes of endpoint analysis. A paired dataset consisted of the commanded threshold and the maximum manual threshold (i.e. the maximum of the manual unipolar and manual bipolar thresholds) obtained at a visit.
Time Frame: 3 months post implant
Population: Pooled subjects with a sufficient pacing output voltage to capture the right atrium at the 1-month and the 3-month follow-up visits.
Measure: Number (95% Confidence Interval); unit: Percentage of RAAT w. sufficient output
Units Other Than Participants: Right Atrial Automatic Threshold Tests
Groups:
- Pooled Pacemaker and CRT-P Population: All Pacemaker implanted subjects and all CRT-P implanted subjects.
Arm/Group | Pooled Pacemaker and CRT-P Population
Number analyzed (Participants) | 132
Number analyzed (Right Atrial Automatic Threshold Tests) | 195
Percentage of RAAT w. sufficient output | 100 [98.5 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Subjects Implanted With a Study Device or Attempted to be Implanted With a Study Device: The study's primary endpoints were designed to assess adverse events for all participants under one category of Cardiac Implantable Electronic Devices (CIED) safety as a unified group. Reporting thus reflects the collective safety profile of CIED interventions as planned and analyzed. This approach was consistent with the study's protocol and objectives, which did not include arm/group-specific AE analysis as a key outcome.
Arm/Group | Subjects Implanted With a Study Device or Attempted to be Implanted With a Study Device
All-Cause Mortality (participants affected / at risk) | 5/136
Serious Adverse Events (participants affected / at risk) | 52/136
Other Adverse Events (participants affected / at risk) | 24/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Subjects Implanted With a Study Device or Attempted to be Implanted With a Study Device (N=136)
PG - Oversensing - RV (Product Issues) | 1 (1)
PG - Infection (> 30 days post-implant) (Product Issues) | 1 (1)
Procedure - Venous occlusion (Vascular disorders) | 2 (2)
Hematoma - Pocket (<=30 days post-implant) (Vascular disorders) | 1 (1)
Renal failure due to contrast media - Procedure (Renal and urinary disorders) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1)
Venous occlusion (Product Issues) | 1 (1)
LV - difficult visualization (Vascular disorders) | 1 (1)
Dislodgment - RA (Product Issues) | 3 (4)
Dislodgment - RV (Product Issues) | 1 (2)
Extracardiac stimulation - LV (Product Issues) | 1/36 (1)
Dyspnea - Heart failure (Cardiac disorders) | 2 (2)
Heart failure symptoms - Unspecified (Cardiac disorders) | 2 (2)
Multiple heart failure symptoms (Cardiac disorders) | 6 (6)
Atrial Arrhythmias (Heart Failure related) (Cardiac disorders) | 1 (1)
Pleural Effusion (Cardiac disorders) | 1 (1)
Atrial fibrillation (AF) (Cardiac disorders) | 5 (5)
Atrial flutter (Cardiac disorders) | 2 (2)
Other SVT (Cardiac disorders) | 1 (1) — AVRT, AVNRT, EAT etc.
Peripheral vascular disease (Vascular disorders) | 2 (3)
Intermittent claudication (Cardiac disorders) | 1 (1)
Aortic regurgitation (Vascular disorders) | 1 (1)
Syncope (Cardiac disorders) | 1 (1)
Dizziness (Cardiac disorders) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1)
Cerebrovascular accident (CVA) (Cardiac disorders) | 1 (1)
Pulmonary embolism (Cardiac disorders) | 1 (1)
Adverse Drug Effect (General disorders) | 1 (2)
Chest Pain (General disorders) | 1 (1)
Multiple symptoms (General disorders) | 1 (1)
Death (Product Issues) | 1 (1)
Death (General disorders) | 1 (1)
Systemic infection (Infections and infestations) | 1 (1)
Physical trauma (Injury, poisoning and procedural complications) | 1 (1)
Hematological (Blood and lymphatic system disorders) | 1 (1)
Neurological (Nervous system disorders) | 2 (2)
Gastrointestinal (Gastrointestinal disorders) | 3 (3)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Genitourinary (Renal and urinary disorders) | 1 (1)
Renal (Renal and urinary disorders) | 4 (6)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (7)
Integumentary (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1 (1)
Immune (Immune system disorders) | 1 (1)
Cancer (General disorders) | 7 (8)
Multi-system failure (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Subjects Implanted With a Study Device or Attempted to be Implanted With a Study Device (N=136)
Extracardiac stimulation - LV (Product Issues) | 11/36 (11) — Extracardiac stimulation - LV, only applicable to LV leads. CRT-P subjects have LV leads implanted, Pacemaker subjects do not have LV leads implanted.
Atrial fibrillation (AF) (Cardiac disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Consultant (PI) acknowledges and agrees that (i) Consultant shall not publish any data, report, white papers or other materials arising out of the Services performed pursuant to this Agreement without the prior written consent of Boston Scientific, and (ii) any such publication shall not include Boston Scientific Confidential Information except prior written consent of Boston Scientific.